CLINICAL TRIAL: NCT06600269
Title: The Effect of Cycling Priming Coordination Training on Ataxia and Brain Plasticity
Brief Title: Cycling-Based Priming Coordination Training for Enhancing Ataxia Recovery and Brain Plasticity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Professor, Chang Gung University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SCA_001
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Spinocerebellar Ataxias
Keywords: Transcranial Magnetic Stimulation (TMS); Gait; Motor Control; Motor Learning
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCA training group (Experimental): Long-term training
  Interventions: Procedure: Cycling Training
- SCA Control group (No Intervention): Control group

INTERVENTIONS:
Procedure: Cycling Training — Cycling combined with priming strategies to enhance motor learning tasks. Each session will last for 15 minutes, conducted three times per week, over a period of two weeks.
  Arms: SCA training group

SUMMARY:
Effective walking and balance require not only lower limb muscle strength but also coordinated movement. For individuals with Spinocerebellar Ataxia (SCA), rehabilitation strategies targeting coordination are essential to improving mobility and reducing the burden on caregivers. However, evidence-based rehabilitation approaches for ataxia remain limited.

Recent studies suggest that improvements in motor learning are often accompanied by changes in cortical excitability. Abnormal cortical excitability in SCA patients may hinder rehabilitation efforts, yet priming strategies-such as exercise or specific stimuli-have been shown to enhance motor learning by modulating cortical excitability. Cycling exercise, in particular, has demonstrated the potential to improve coordination and influence cortical plasticity in individuals with SCA, making it a promising priming strategy for coordination training.

This clinical trial aims to:

1. Investigate the priming effect and neural mechanisms of acute cycling exercise on coordination training in patients with SCA.
2. Explore the long-term impact of priming cycling training on cortical plasticity and functional mobility in individuals with SCA.

This study seeks to provide insights into optimized rehabilitation interventions that could enhance the quality of life and independence for people with SCA.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of SCA.

Exclusion Criteria:

* Musculoskeletal injuries on legs
* Osteoporosis.
* Any peripheral or central nervous system injury or disease patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-04 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Overall Response Time | Baseline, 2 weeks and 4 weeks
  The sum of reaction time and movement time, providing a complete measure of the time taken from the stimulus presentation to the completion of the response. Unit: Second(s)
Overall Error Rate | Baseline, 2 weeks and 4 weeks
  The total proportion of incorrect responses across a testing session or series of tasks.
Motor Evoked Potentials (MEPs) | Baseline, 2 weeks and 4 weeks
  MEPs are the electrical responses recorded from muscles following stimulation of the motor cortex. They reflect the efficiency of neural transmission from the cortex to the muscle. Unit: millivolts (mV).
Intracortical Facilitation (ICF) | Baseline, 2 weeks and 4 weeks
  ICF is measured by applying a pair of TMS pulses with a short interval (e.g., 8-15 ms) where the first (subthreshold) pulse is followed by a second (suprathreshold) pulse, leading to an increased amplitude of the MEP.
Intracortical Inhibition (ICI) | Baseline, 2 weeks, and 4 weeks
  ICI is measured similarly to ICF but with a shorter inter-stimulus interval (e.g., 1-5 ms), resulting in a suppressed MEP amplitude. This suppression reflects inhibitory processes within the cortex.
Total Scale for the Assessment and Rating of Ataxia (SARA) Score | Baseline, 2 weeks, and 4 weeks
  To objectively assess ataxia severity across various domains of motor function including gait, stance, sitting, speech disturbance, finger chase, nose-finger test, fast alternating hand movements, and heel-shin slide. Each item is scored individually with a scale that typically ranges from 0 (no ataxia) to a maximum score that depends on the severity and the aspect of ataxia being assessed. The total score ranges from 0 (no ataxia) to 40 (most severe ataxia).
Total Berg Balance Scale (BBS) Score | Baseline, 2 weeks, and 4 weeks
  To measure an individual's balance abilities through various tasks that mimic daily activities, assessing the risk of falls and overall balance proficiency. The BBS consists of 14 items that evaluate a range of functions including sitting to standing, standing unsupported, transferring, turning to look behind, picking up an object from the floor, and standing on one leg. Each task is rated on a scale from 0 (unable) to 4 (independent), with the total score ranging from 0 to 56. A higher total score indicates better balance and lower fall risk. Scores below 45 are generally indicative of increased fall risk.
Total Time to Complete the Time Up and Go test (TUG test) | Baseline, 2 weeks, and 4 weeks
  The time, in seconds, it takes for a participant to complete the TUG test from the initial sitting position to returning to the seated position. An older adult who takes ≥12 seconds to complete the TUG is at risk for falling.
Walking Speed | Baseline, 2 weeks, and 4 weeks
  The time taken by participants to walk a standardized distance, typically expressed in centimeters per second (cm/s).
Step Length | Baseline, 2 weeks, and 4 weeks
  The linear distance between the two ankles, typically expressed in centimeter(cm).
Step Time | Baseline, 2 weeks, and 4 weeks
  The duration taken for one complete step, measuring from foot-off of one foot to the next foot-off of the same foot, usually expressed in seconds.
Fatigue Level Measurement Using Multidimensional Fatigue Inventory (MFI) | Baseline, 2 weeks, and 4 weeks
  The MFI is a 20-item self-report questionnaire used to measure five dimensions of fatigue: general fatigue, physical fatigue, mental fatigue, reduced activity, and reduced motivation. Each dimension is scored separately, with higher scores indicating greater fatigue
Sleep Quality Measurement Using Pittsburgh Sleep Quality Index (PSQI) | Baseline, 2 weeks, and 4 weeks
  The PSQI is a 19-item self-report questionnaire that assesses sleep quality over a 1-month period. It generates a global score ranging from 0 to 21, with higher scores indicating poorer sleep quality. The PSQI includes seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction.

SECONDARY OUTCOMES:
Gait Speed Measurement Using 10-Meter Walk Test (10MWT) | Baseline, 2 weeks, and 4 weeks
  The 10MWT is a performance-based measure used to assess walking speed over a short distance. Participants will be instructed to walk 10 meters at their comfortable and/or fastest walking speed. The time taken to walk the central 6 meters is recorded to eliminate acceleration and deceleration effects, and gait speed is calculated as meters per second (m/s).
Double Support Time | Baseline, 2 weeks, and 4 weeks
  The portion of the gait cycle where both feet are in contact with the ground, indicating the transition phase between steps, expressed as a percentage of the gait cycle or in seconds.
Single Support Time | Baseline, 2 weeks, and 4 weeks
  The duration within the gait cycle when only one foot is in contact with the ground, typically measured in seconds or as a percentage of the total gait cycle.
Swing Time | Baseline, 2 weeks, and 4 weeks
  The portion of the gait cycle where the foot is not in contact with the ground, moving forward to the next step. It is usually expressed as a percentage of the total gait cycle or in seconds.
Stance Time | Baseline, 2 weeks, and 4 weeks
  The portion of the gait cycle when the foot is in contact with the ground, supporting body weight. It's typically expressed as a percentage of the total gait cycle or in seconds
Cadence | Baseline, 2 weeks, and 4 weeks
  The number of steps an individual takes per minute, providing an overview of gait speed and rhythm, , expressed as steps per minute.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan